CLINICAL TRIAL: NCT04340024
Title: Discovery of Biomarkers for Intrinsic Radiation Sensitivity in Cancer Patients
Status: Recruiting | Type: Observational
Sponsor: National Cancer Centre, Singapore (Other)
Collaborators: National Medical Research Council (NMRC), Singapore (Other Government); Duke-NUS Graduate Medical School (Other); Ferring Pharmaceuticals (Industry); ImmunoSCAPE (Industry); Decipher Biosciences (Unknown)
Responsible Party: Sponsor
Other Study IDs: DISCLOSE
Record Dates: First submitted 2020-03-26; First posted 2020-04-09 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Nasopharyngeal Cancer; Prostate Cancer; Other Cancer
Keywords: Radiotherapy; Biomarkers; Genomics; Immunomics; Precision medicine
MeSH Terms: conditions — Nasopharyngeal Neoplasms; Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — 20mL of blood will be collected up to 5 times over 5 years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients with cancers that are sensitive to radiotherapy treatment and/or patients who have experienced severe acute/ late side effects to radiotherapy will be recruited to the study. Blood and/or matched tumour-normal tissue pairs will be collected. Blood and/or tissue samples will be processed and studied for genetic and biochemical markers that have potential to be used for predicting sensitivity to radiation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with severe side effects from radiotherapy
* Patients with a type of cancer that is associated with sensitivity to radiotherapy

Exclusion Criteria:

* Age of patient must be between 21 (inclusive) and 99 (exclusive)

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from patients of the study team when they attend their regular clinic visits or when they are admitted to the hospital. These are patients from NCCS.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2015-09-30 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
To identify genes or molecular pathways that are associated with radiation sensitivity in blood and tissue samples | Blood is taken at informed consent; tissue is from archived sample
  Whole exome sequencing, single nucleotide polymorphism (SNP) assays
Change in immune profile of blood and tissue after radiation | Blood is taken at informed consent; tissue is from archived sample
  Mass cytometry using CyTOF technology will be used to detect the immune cell population
To identify proteins that are associated with radiation sensitivity in tissue samples | Tissue is from archived sample
  Immunohistochemistry will be used to detect protein expression
To identify RNA expression pathways that are associated with radiation sensitivity in blood and tissue samples | Blood is taken at informed consent; tissue is from archived sample
  RNA sequencing

CONTACTS AND LOCATIONS:
Overall Officials: Melvin Chua, MD, Principal Investigator — National Cancer Centre, Singapore
Locations (1):
- National Cancer Center Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No